CLINICAL TRIAL: NCT03262168
Title: Supported Exercise Programme for Adults With Congenital Heart Disease (SEA CHange)
Brief Title: Supported Exercise Programme for Adults With Congenital Heart Disease
Acronym: SEACHange
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Golden Jubilee National Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GoldenJNH
Record Dates: First submitted 2017-04-07; First posted 2017-08-25 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Congenital Disorder; Heart Diseases
Keywords: Exercise; Physical Activity
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Heart Diseases; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants compete a six minute walk test (6MWT). Those who achieve less than 450 metres will be assigned to study group one. Participants who achieve greater than 450 metres on 6MWT will be assigned to study group two.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Study Group One (Other): Six Minute Walk Test distance <450metres. Exercise programme including inspiratory muscle trainer for 12 weeks. Contact weekly (via phone or email).
  Interventions: Other: Exercise Programme
- Study Group Two (Other): Six Minute Walk Test distance >450metres. Exercise programme including walking for 12 weeks. Contact every second week (via phone or email).
  Interventions: Other: Exercise Programme
- Study Group One - phase 2 (Other): Six Minute Walk Test distance <450metres. Exercise programme including inspiratory muscle trainer for 12 weeks. Contact weekly (via phone or email).
  Interventions: Other: Exercise Programme
- Study Group Two - phase 2 (Other): Six Minute Walk Test distance >450metres. Exercise programme including walking for 12 weeks. Contact every second week (via phone or email).
  Interventions: Other: Exercise Programme

INTERVENTIONS:
Other: Exercise Programme — Complete background demographics, Sniff Nasal Inspiratory Pressure (study group one only), grip strength, muscle strength, PHQ-9 and GAD-7 questionnaires.

SUMMARY:
This study will evaluate if the introduction of a supported exercise programme can improve physical and psychological well-being for adults with congenital heart disease.

DETAILED DESCRIPTION:
Congenital heart disease (CHD) describes heart defects present from birth. The majority of affected patients will require lifelong care to not only manage their medical condition, but also to offer support and guidance on living with their specific heart condition. Exercise and physical activity is one such area where patients often require support and advice. Recommendations are in place for health care providers to promote physical activity for this patient population. However, many health care providers find it difficult to know what level of exercise is reasonable or how to escalate current exercise programmes.

The benefits of regular exercise are well known and evidence suggests that even a modest increase in physical activity can reduce morbidity, improve psychological wellbeing and protect against cardiovascular disease.

This pilot study will determine the feasibility of introducing a supported exercise programme to clinical practice. The investigators aim to assess if improvements can be made in both physical and psychological well-being for adults with CHD who are living in Scotland. After initial assessment and baseline measurements are obtained, participants will follow a twelve week individualised programme. The investigators will keep in regular contact with the participant throughout and arrange interval and final assessments. The baseline measurements will be repeated during the final assessment at 12 weeks. Investigators anticipate that the study will also help to establish a programme that will help to improve the way adults who were born with a heart condition can be supported with physical activity on a long term basis.

ELIGIBILITY:
Inclusion Criteria:

* Living in Scotland
* Diagnosis of congenital heart disease
* Walks less than 450 metres on a 6 minute walk test (Group 1)
* Walks more than 450 metres on a 6 minute walk test (Group 2)

Exclusion Criteria:

* No access to internet or telephone
* Non English speaking (If the pilot study is successful, we anticipate that materials and programmes could be translated and accessible to non English speakers)
* Vulnerable adults
* Severe aortic stenosis or severe left ventricular outflow tract obstruction (LVOTO)
* Eisenmenger Physiology (ongoing study recruitment with SPVU)
* Currently prescribed Advanced Pulmonary Vasodilator therapy

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Attendance rate | 12 weeks (for each phase)
  Determine the feasibility of introducing a supported exercise programme in to clinical practice. This will be measured through attendance to the programme and interaction with the online resource.
Attrition rate | 12 weeks (for each phase)
  Determine the feasibility of introducing a supported exercise programme by assessing attrition rate throughout the study period.

SECONDARY OUTCOMES:
Change in six minute walk test (6MWT) | 12 weeks (for each phase)
  Change in six minute walk test distance (metres) between 0 and 12 weeks. Offers a simple, readily available and cost effective method for objective evaluation of functional exercise capacity during daily activity.
Change in Sniff Nasal Inspiratory Pressure (SNIP) | 12 weeks (for each phase)
  Change in Sniff Nasal Inspiratory Pressure (SNIP) between 0 and 12 weeks (study group one). Measured in cmH2O and is used to measure inspiratory muscle strength.
Change in Grip Strength | 12 weeks (for each phase)
  Change in grip strength. This is measured in pounds (lbs) using a myometer. It is a recognized method of assessing overall nutritional status and health in subjects with medical conditions.
Is there an improvement in level of psychological distress | 12 weeks (for each phase)
  Change in level of depression (measured using PHQ- 9 questionnaire). It is a reliable and validated self report questionnaire used to help clinicians screen for depression disorder.
Is there an improvement in level of psychological distress | 12 weeks (for each phase)
  Change in level of anxiety (measured using GAD-7 questionnaire). The GAD -7 is a self report questionnaire used to identify probable cases of generalised anxiety disorder. Recognised as a valid and reliable screening tool
Body mass Index (BMI) | 12 weeks (for each phase)
  Change in body mass index (measured in kg/m2). Weight (kgs) and height (metres) will be combined to report BMI in kg/m2
Body weight | 12 weeks (for each phase)
  Change in body weight (measured in kg)
Is there an improvement in bicep strength | 12 weeks (for each phase)
  Change in bicep strength. This is measured in newtons (N) using a non invasive strain guage/myometer
Is there an improvement in quadricep strength | 12 weeks (for each phase)
  Change in quadricep strength. This is measured in newtons (N) using a non invasive strain guage/myometer

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Mason, MSc, Study Chair — Golden Jubilee Research Institute
Locations (1):
- Golden Jubilee National Hospital, Clydebank, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share individual data